CLINICAL TRIAL: NCT00750308
Title: Renin Angiotensin Aldosterone System (RAAS) and Fibrinolysis in Humans: ACEi
Brief Title: Renin Angiotensin Aldosterone System (RAAS) and Fibrinolysis in Humans: ACEi and PE5i
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 060198
Record Dates: First submitted 2008-09-05; First posted 2008-09-10 (Estimated); Results first posted 2010-04-12 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Ramipril; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- tadalafil, ramapril, combo, placebo (Active Comparator): placebo+tadalafil for three weeks, washout, placebo+ramipril for three weeks, washout, ramipril + tadalafil, washout, placebo+placebo for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- ramipril, tadalafil, placebo, combo (Active Comparator): placebo+ramipril for three weeks, washout, placebo+tadalafil for three weeks, washout, placebo+placebo for three weeks, washout, ramipril+tadalafil for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- combo, placebo, tadalafil, ramipril (Active Comparator): ramipril+tadalafil for three weeks, washout, placebo+placebo for three weeks, washout, placebo+tadalafil for three weeks, washout, placebo+ramipril for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- placebo, combo, ramipril, tadalafil (Active Comparator): placebo+placebo for three weeks, washout, ramipril+tadalafil for three weeks, washout placebo+ramipril for three weeks, washout, placebo+tadalafil for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- tadalafil, placebo, ramipril, combo (Active Comparator): placebo+tadalafil for three weeks, washout, placebo+placebo for three weeks, washout, placebo+ramipril for three weeks, washout, ramipril+tadalafil for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- ramipril, combo, tadalfil, placebo (Active Comparator): placebo+ramipril for three weeks, washout, ramipril+tadalafil for three weeks, washout, placebo+tadalafil for three weeks, washout, placebo for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- combo, ramipril, placebo, tadalafil (Active Comparator): ramipril+tadalafil for three weeks, washout, placebo+ramipril for three weeks, washout, placebo+placebo for three weeks, washout, placebo+tadalafil for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- placebo, tadalafil, combo, ramipril (Active Comparator): placebo+placebo for three weeks, washout, placebo+tadalafil for three weeks, washout, ramipril+tadalafil for three weeks, washout, placebo+ramipril for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- tadalafil, combo, placebo, ramipril (Active Comparator): placebo+tadalafil for three weeks, washout, ramipril+tadalafil for three weeks, washout, placebo+placebo for three weeks, washout, placebo+ramipril for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- ramipril, placebo, combo, tadalafil (Active Comparator): placebo+ramipril for three weeks, washout, placebo+placebo for three weeks, washout, ramipril+tadalafil for three weeks, washout, placebo+tadalafil for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- combo, tadalafil, ramipril, placebo (Active Comparator): ramipril+tadalafil for three weeks, washout, placebo+tadalafil for three weeks, washout, placebo+ramipril for three weeks, washout, placebo+placebo for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo
- placebo, ramipril, tadalafil, combo (Active Comparator): placebo+placebo for three weeks, washout, placebo+ramipril for three weeks, washout, placebo+tadalafil for three weeks, washout, ramipril+tadalafil for three weeks
  Interventions: Drug: Ramipril; Drug: Tadalafil; Drug: placebo

INTERVENTIONS:
Drug: Ramipril — Ramipril 10 mg per day for three weeks
  Other Names: Altace
Drug: Tadalafil — tadalafil 10 mg every other day for three weeks
  Other Names: Cialis
Drug: placebo — placebo matching ramipril
  Other Names: matching ramipril
Drug: placebo — placebo matching tadalafil
  Other Names: matching tadalfil

SUMMARY:
This study will measure the effect of the agent tadalafil on glucose and insulin homeostasis in people with metabolic syndrome in the presence and absence of an ACE inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects, 18 to 70 years of age, inclusive
2. For female subjects, the following conditions must be met:

   * Postmenopausal status for at least 1 year,
   * Status-post surgical sterilization, or
   * If of childbearing potential, utilization of adequate birth control, and willingness to undergo urine beta-hcg testing prior to drug treatment and on every study day
3. Metabolic syndrome as defined by 3 or more of the following:

   * Fasting plasma glucose of at least 100 mg/dL (5.5 mmol/L),
   * Serum triglycerides of at least 150 mg/dL (1.7 mmol/L),
   * Serum HDL cholesterol less than 40 mg/dL (1.04 mmol/L) in males and less than 50mg/dl (1.30mmol/L) in females,
   * Blood pressure of at least 130/85 mmHg, or
   * Waist girth of more than 102 cm in men or 88 cm in women

Exclusion criteria:

Subjects presenting with any of the following will not be included in the study:

1. Diabetes type 1 or type 2, as defined by a fasting glucose of 126 mg/dL or greater or the use of anti-diabetic medication
2. Use of hormone replacement therapy
3. Statin therapy
4. In hypertensive subjects, a seated systolic blood pressure greater than 179 mmHg or a seated diastolic blood pressure greater than 110 mmHg
5. Pregnancy
6. Breast-feeding
7. Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
8. Treatment with anticoagulants
9. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
10. History or presence of immunological or hematological disorders
11. Diagnosis of asthma
12. Clinically significant gastrointestinal impairment that could interfere with drug absorption
13. Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] > 1.5 x upper limit of normal range)
14. Impaired renal function (serum creatinine > 1.5 mg/dl)
15. Hematocrit < 35%
16. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
17. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
18. Treatment with lithium salts
19. History of alcohol or drug abuse
20. Treatment with any investigational drug in the 1 month preceding the study
21. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
22. Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, M.D., Principal Investigator — Vanderbilt University Medical Center

RESULTS

PARTICIPANT FLOW:
Period: First Treatment
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 (One female withdrew due to muscle pain) | 3 | 2 | 2 | 2 | 3 | 2 | 3 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 1 | 2 | 3 | 2 | 2 | 2 | 2 | 1 | 1
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 | 2 | 2 | 1 | 2 | 3 | 2 | 2 | 2 | 2 | 1 | 1
Completed | 2 | 2 | 2 | 1 | 2 | 3 | 2 | 2 | 2 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Treatment
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 | 2 | 2 | 1 | 2 | 3 | 2 | 2 | 2 | 2 | 1 | 1
Completed | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Completed | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Treatment
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Completed | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Completed | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Treatment
Arm/Group | Tadalafil, Ramipril, Combo, Placebo | Ramipril, Tadalafil, Placebo, Combo | Combo, Placebo, Tadalafil, Ramipril | Placebo, Combo, Ramipril, Tadalafil | Tadalafil, Placebo, Ramipril, Combo | Ramipril, Combo, Tadalafil, Placebo | Combo, Ramipril, Placebo, Tadalafil | Placebo, Tadalafil, Combo, Ramipril | Tadalafil, Combo, Placebo, Ramipril | Ramipril, Placebo, Combo, Tadalafil | Combo, Tadalafil, Ramipril, Placebo | Placebo, Ramipril, Tadalafil, Combo
Started | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Completed | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We provide baseline data for those 18 subjects who completed all four treatment arms and whose data are analyzed in this crossover study.
Groups:
- Completed Subjects: Subjects who completed all four treatment arms.
Arm/Group | Completed Subjects
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Beta Cell Function
Description: Beta cell function as measured during a frequently sampled IV glucose tolerance test
Time Frame: 3 hours
Measure: Mean (Standard Error); unit: microU/mM
Groups:
- Placeb Treatment: Measurements during placebo treatment for all 18 subjects who completed the protocol
- Ramipril Treatment: Measurements during ramipril treatment for all 18 subjects who completed the protocol
- Tadalafil Treatment: Measurements during tadalafil treatment for all 18 subjects who completed the protocol
- Combination Treatment: Measurements during combination (ramipril and tadalafil) for all 18 subjects who completed the protocol
Arm/Group | Placeb Treatment | Ramipril Treatment | Tadalafil Treatment | Combination Treatment
Number analyzed (Participants) | 18 | 18 | 18 | 18
microU/mM | 241.2 (45.2) | 232.3 (38.1) | 292.1 (38.9) | 287.6 (54.3)

2. Primary Outcome: Insulin Sensitivity
Description: As assessed using IV glucose tolerance test and calculated using Min Mod units mU/mm
Time Frame: three weeks
Population: Those who completed protocol
Measure: Mean (Standard Error); unit: (mU/L)-1x(min)-1xL
Groups:
- Placebo Treatment: Measured during placebo treatment in all 18 subjects who completed the study
- Ramipril Treatment: Measured during ramipril treatment in all 18 subjects who completed the protocol
- Tadalafil Treatment: Measured during tadalafil in all 18 subjects who completed the protocol
- Combination Treatment: Measured during combination (ramipril and tadalafil) in all 18 subjects who completed treatment
Arm/Group | Placebo Treatment | Ramipril Treatment | Tadalafil Treatment | Combination Treatment
Number analyzed (Participants) | 18 | 18 | 18 | 18
(mU/L)-1x(min)-1xL | 2.21 (0.35) | 1.76 (0.34) | 1.88 (0.25) | 1.76 (0.29)

ADVERSE EVENTS:
Groups:
- Placebo Treatment: Any adverse event that occurred during placebo treatment in anyone who received placebo treatment
- Ramipril Treatment: Any adverse event that occured durng ramipril treatment in anyone who received ramipril treatment
- Tadalafil Tretament: Any adverse event that occurred during tadalafil treatment in anyone who received tadalafil treatment
- Combination Treatment: Any adverse event that occurred during combination (ramipril and tadalafil) treatment in anyone who received combination treatment
Arm/Group | Placebo Treatment | Ramipril Treatment | Tadalafil Tretament | Combination Treatment
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 1/23 | 3/24 | 0/23 | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment (N=23) | Ramipril Treatment (N=24) | Tadalafil Tretament (N=23) | Combination Treatment (N=25)
muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No